CLINICAL TRIAL: NCT03095183
Title: Do Traditional or Flavored Tongue Depressors Make for Easier Posterior
Brief Title: Do Traditional or Flavored Tongue Depressors Make for Easier Posterior Oropharynx Exams in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian P. Murray, DO, Senior Resident, Emergency Medicine, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: C.2016.146d
Record Dates: First submitted 2017-02-27; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Oropharynx
Keywords: Posterior oropharynx exam; Pediatric; Tongue Depressor; Flavored Tongue Depressor

STUDY DESIGN:
Intervention Model Description: All patients registered for evaluation in the Brooke Army Medical Center Pediatric Emergency Department will be screened by evaluation of age, mental status, physical features and history of immunocompromised by the PI or AI as part of their standard triage and care procedures for their evaluation and treatment in the Emergency Department. Potential participants will be identified by the PI and AI from patients who are registered to be seen by the PI or AI. Potential participants who meet the inclusion criteria and who have none of the exclusion criteria will be approached prior to completion of the posterior oropharynx exam for permission to enroll them in this study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Using a computer-generated simple randomization sequence in permuted blocks of 10, numbered study packets that include the surveys and tongue depressor will be prepared in advance. The packets, which will be prepared by a third party not participating in this research study, will include the information sheet, surveys for the investigator, participant and parent, all labeled with the sample number, and a tongue depressor within original packaging. The randomization key will be kept by the third party until the completion of data collection, at which time it will be given to the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional Tongue Depressor (Placebo Comparator): The posterior oropharynx exam was performed with a traditional, unflavored Puritan Regular tongue depressor.
  Interventions: Device: Traditional unflavored Puritan Regular Tongue Depressor
- Flavored Tongue Depressor (Active Comparator): The posterior oropharynx exam was performed with a grape flavored, commercially available, Puritan Junior tongue depressor.
  Interventions: Device: Grape flavored Puritan Junior tongue depressor

INTERVENTIONS:
Device: Grape flavored Puritan Junior tongue depressor
  Arms: Flavored Tongue Depressor
Device: Traditional unflavored Puritan Regular Tongue Depressor
  Arms: Traditional Tongue Depressor

SUMMARY:
Evaluation of the oropharynx is a standard component of a general medical exam for all pediatric patients, but is an essential exam in the undifferentiated ill child. Pediatric patients are unable to verbalize where they hurt, and a comprehensive evaluation is needed to identify the source of fever and illness. Frequently, illnesses will present atypically as well, and a patient complaining of abdominal pain may ultimately be diagnosed with streptococcus pharyngitis. If the examiner does not evaluate the posterior oropharynx, the throat as a cause of abdominal pain is easily overlooked. Additionally, young children are prone to infections with pox viruses causing herpangina, hand foot and mouth disease, oral thrush. Despite the importance of the posterior oropharynx exam, it can be a source of stress and anxiety for both the clinician and pediatric patient when a tongue depressor is used to evaluate the posterior oropharynx. However, there are no studies to date that have looked at decreasing the difficulty or at decreasing the perceived discomfort associated with the poster oropharynx exam in the pediatric patient when a tongue depressor is utilized. Despite this paucity of research, there are multiple different flavored and candied tongue depressors available for this purpose which may or may not aid in obtaining posterior oropharynx exam and decrease the discomfort experienced by the patients.

DETAILED DESCRIPTION:
The study design is a prospective, placebo-controlled, randomized controlled trial using a convenience sample of 96 pediatric patients presenting for care in the emergency department who require an oropharyngeal examination as part of their evaluation. Examinations will be performed utilizing either traditional (unflavored) or flavored tongue depressors in a random fashion. . Physician/provider investigators will complete a brief survey after each exam as to the ease of the exam and the perceived emotional discomfort the exam experienced by the subject, both recorded on a visual analog scale. The age and sex of the subject, and the education level of the investigator will also be recorded. A single question survey will also be provided to the parent/caregiver as to their perception of the discomfort of their child during the posterior oropharynx exam using a visual analog scale. Additionally, a single question survey will be posed to the subject asking for their discomfort level during the exam using the Oucher pediatric pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 3 and 12 years of age presenting to the emergency department who require the use of a tongue depressor to evaluate the posterior pharynx as part of their clinical evaluation.

Exclusion Criteria:

* Patients who do not require a tongue depressor to fully examine the posterior oropharynx, patients who are immunocompromised and patients who are younger than 3 years of age or older than 12 years of age. We will also exclude patients with abnormal facies, and any patients with altered mental consciousness as defined by a GCS less than 15.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Does the use of a flavored tongue depressor decrease the patient's actual discomfort during a posterior oropharynx exam using the Oucher pediatric pain scale? | Up to 12 months

SECONDARY OUTCOMES:
Do flavored tongue depressors increase the ease of the posterior oropharynx exam in the pediatric patient by provider subjective assessment? | Up to 12 months
Does the use of a flavored tongue depressor decrease the perceived discomfort associated with pediatric posterior oropharynx exam as determined by the provider subjective assessment? | Up to 12 months
Does the use of a flavored tongue depressor decrease the perceived discomfort associated with pediatric posterior oropharynx exam as determined by the patient's caregiver? | Up to 12 months

IPD SHARING:
Plan to Share IPD: Undecided